CLINICAL TRIAL: NCT05232240
Title: Blood Pressure Variability in Non-hypertensive Patients With Ischemic Cerebrovascular Disease
Acronym: BPV-NhICVD
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xin Ma, Principal investigator, Xuanwu Hospital, Beijing
Other Study IDs: BPV-NhICVD
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Ischemic Cerebrovascular Disease; Blood Pressure Variability
Keywords: ischemic stroke; transient ischemic attack; non-hypertensive; blood pressure variability; vascular risk
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-hypertensive patients with Ischemic Cerebrovascular Disease: The patients are diagnosed as ischemic cerebrovascular disease (ICVD) and less than 90 days after the onset of ischemic stroke or transient ischemic attack. The patients have no definite diagnosis of hypertension, and are not under anti-hypertension treatment. The blood pressure measured 5~90 days after the ICVD onset without any anti-hypertension treatment is less than 140/90 mmHg (an average of ≥ 2 readings obtained on ≥ 2 occasions after emptying bladder, relaxing for more than 5 min, and avoiding caffeine, exercise, or smoking for at least 30 min before measurement).
  Interventions: Diagnostic Test: blood pressure variability measured by ambulatory 24-hour blood pressure monitoring

INTERVENTIONS:
Diagnostic Test: blood pressure variability measured by ambulatory 24-hour blood pressure monitoring — The ambulatory 24-hour blood pressure monitoring will be performed at baseline and one year after the enrollment. Various blood pressure variability characteristics will be obtained from these examinations.

SUMMARY:
This study is a single-center prospective cohort of patients with ischemic cerebrovascular disease (ICVD) who have not met the diagnostic criteria for hypertension. Ambulatory 24-hour blood pressure monitoring (ABPM) will be performed at baseline and one year after the enrollment. The primary purpose of the study is to delineate the relationship of blood pressure variability (BPV) with the risk of composite vascular events in non-hypertensive patients with ICVD. The factors related to BPV, as well as the potential modulators of the associations between BPV and vascular risk, will be further explored among these patients.

DETAILED DESCRIPTION:
Hypertension is one of the most important risk factors of ischemic cerebrovascular disease (ICVD), while various blood pressure variability (BPV) indices are immerging as novel prognostic indicators independent of the blood pressure level. However, the BPV profiles without hypertension have not been specifically observed. Considering the great importance of blood pressure management in ICVD, more research is needed to clarify whether and how BPV will increase the vascular risk in non-hypertensive patients with ICVD. This prospective cohort study will be helpful to invoke an early management of blood pressure in patients with ICVD before the clinical establishment of hypertension.

All eligible non-hypertensive patients hospitalized for ICVD will be consecutively enrolled in this cohort. Blood pressure measurements are obtained with ambulatory 24-hour blood pressure monitoring (ABPM) every 20 minutes during day-time (6:00-22:00) and every 30 minutes during night-time (22:00-6:00) at baseline and one year after the enrollment. The clinical, imaging and laboratory information will be collected at baseline. During an estimated 3-year follow-up, the vessel-related diagnostic or monitoring procedures, treatment, functional status and new vascular events will be recorded by web-based patients' self-reports and investigators' regular telephone visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as ischemic stroke or transient ischemic attack (TIA), with confirmation of computed tomography or magnetic resonance imaging.
2. Less than 90 days after onset of ischemic stroke or TIA symptoms.
3. The blood pressure measured 5~90 days after the ICVD onset without any anti-hypertension treatment is less than 140/90 mmHg (an average of ≥2 readings obtained on ≥ 2 occasions after emptying bladder, relaxing for more than 5 min, and avoiding caffeine, exercise, or smoking for at least 30 min before measurement).
4. Consent to participate in the study.

Exclusion Criteria:

1. A definite diagnosis of hypertension.
2. Under anti-hypertension treatment.
3. Worsening neurological conditions.
4. With a National Institute of Health Stroke Scale score more than 5 points.
5. Intracranial hemorrhage.
6. Autonomic failure.
7. With malignant tumors or poor organ functions or hematologic diseases, whose estimated life expectancy is less than 3 years.
8. With contraindications to ambulatory 24-hour blood pressure monitoring or fail to finish the examination at baseline.
9. Mental disease.
10. Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are diagnosed as ischemic cerebrovascular disease (ICVD) and less than 90 days after the onset of ischemic stroke or transient ischemic attack. The patients have no definite diagnosis of hypertension, and are not under anti-hypertension treatment. The blood pressure measured 5~90 days after the ICVD onset without any anti-hypertension treatment is less than 140/90 mmHg (an average of ≥ 2 readings obtained on ≥ 2 occasions after emptying bladder, relaxing for more than 5 min, and avoiding caffeine, exercise, or smoking for at least 30 min before measurement).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
3-year risk of Major Adverse Cardiovascular Event | 3 years
  the time of first documented cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction or unstable angina

SECONDARY OUTCOMES:
90-day Functional Outcome | 90 days
  percentage of patients with modified Rankin Scale (mRS) scores (minimum 0 and maximum 5) 3 to 5, who are considered to be disabled
1-year rate of Major Adverse Cardiovascular Event | 1 year
  the rate of cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, and unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina
1-year rate of Ischemic Stroke | 1 year
  the rate of fatal and nonfatal ischemic stroke
1-year rate of Acute Coronary Syndrome | 1 year
  the rate of first documented fatal and nonfatal myocardial infarction and unstable angina
1-year rate of Cardiovascular Mortality | 1 year
  the rate of mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, and unobserved sudden death
3-year risk of Ischemic Stroke | 3 years
  the time of first documented fatal or nonfatal ischemic stroke
3-year risk of Acute Coronary Syndrome | 3 years
  the time of first documented fatal or nonfatal myocardial infarction or unstable angina
3-year risk of Cardiovascular Mortality | 3 years
  the time of mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, BJ, China